CLINICAL TRIAL: NCT02842554
Title: Training "Pain Connoisseurs" for Efficient Analgesic Proof-of-Concept Studies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Analgesic Solutions (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: GRN.PC.002
Record Dates: First submitted 2013-08-21; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Painful Diabetic Neuropathy (PDN)
Keywords: PDN; Painful Diabetic Neuropathy; Diabetes
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- DPA (Other): Drug Placebo Administration
  Interventions: Drug: Drug Placebo Administration
- C (Other): Control
  Interventions: Other: C
- EPT (Other): Evoked Pain Training
  Interventions: Other: EPT

INTERVENTIONS:
Other: EPT
  Arms: EPT
Drug: Drug Placebo Administration
  Arms: DPA
Other: C — No Intervention
  Other Names: Control
  Arms: C

SUMMARY:
The purpose of this study is to assess the ability of Evoked Pain Training (EPT) and Drug/ Placebo Administration (DPA) training to increase subjects' ability to discriminate between active and placebo treatments in a double-blind crossover trial of a known analgesic, measured by standardized effect size, relative to untrained control subjects.

ELIGIBILITY:
Inclusion criteria:

A subject must meet all of the following criteria to be enrolled in the study:

1. Be a man or a non-pregnant, non-lactating woman 18 years or older. Women of childbearing potential should be willing to use an acceptable birth control method (at the Investigator's discretion) during the study to avoid pregnancy.
2. Have voluntarily provided written informed consent.
3. Be able to speak, read, write, and understand English, understand the consent form, complete study-related procedures, and communicate with the study staff.
4. Have a clinical diagnosis of Painful Diabetic Neuropathy (PDN) for at least 6 months.

   a. Clinical diagnosis may be verified by medical records or by clinical examination during the first visit combined with a medical history of appropriate symptoms for at least 6 months.
5. Have a pain intensity score averaging ≥4 on a 0-10 NRS for average daily recall over past 24 hours. (This applies at V1, V2, and V5.)
6. Have an average daily pain intensity of at least 4 on the 0-10 NRS on at least 20 out of the past 30 days.
7. Be, in the opinion of the Investigator, in sufficiently good health to participate in the study at screening, based upon the results of a medical history, physical examination and laboratory analysis.

Prior to each Treatment Period, the participants must meet the following additional criteria for randomization: Have average pain intensity (24-hour recall) ≥4 on the 0-10 NRS.

Exclusion criteria:

A subject must be excluded if any of the following criteria are met:

1. Are pregnant and/or lactating.
2. Have been diagnosed as having any inflammatory arthritis, gout, pseudo-gout, Paget's disease, fibromyalgia or any chronic pain syndrome that in the Investigator's opinion would interfere with the assessment or self-evaluation of pain and other symptoms of PDN.
3. Have evidence for multiple causes of pain in the neuropathic pain area, such as lumbar radiculopathy.
4. Have received or used any of the excluded/prohibited treatments or drugs specified in the list of prohibited treatments (below) or are unable to agree to the list of treatments prohibited during the study.
5. Have a history of congestive heart failure, unstable coronary artery disease, stroke, or uncontrolled hypertension.
6. Have a history of significant gastrointestinal disease, including active gastro-duodenal ulcerations, perforations, or bleeds.
7. Have abnormal clinical laboratory test results or vital signs unless deemed not clinically significant by the investigator.
8. Have regularly worn false fingernails within the past 6 months (more than 25% of the time)
9. Are undergoing active treatment for cancer, are known to be infected by human immunodeficiency virus, or are being acutely and intensively immunosuppressed following transplantation.
10. Have a history of alcohol or other substance abuse (not including nicotine or tobacco) within 5 years.
11. Have a history of suicide attempt within the past 1 year or suicidal ideation within the past 1 month.
12. Have a history of epilepsy or other seizure disorder.
13. Have creatinine clearance below 60 mL/min as calculated by Cockroft-Gault equation for serum creatinine.
14. Known to have a condition that in the Investigator's judgment precludes participation in the study.
15. Have previously been admitted to this study.
16. Are involved in a worker's compensation, disability claim, or litigation related to medical condition or treatment that is open or was settled within the past 12 months. (Whether litigation is related to medical condition or treatment may be decided at the Investigator's discretion. Claims settled >12 months previously are permitted.)
17. Have a known failure to respond to pregabalin, gabapentin, or oxycodone due to either efficacy or tolerability in previous treatment at therapeutically appropriate doses.
18. Are allergic to or have a hypersensitivity to pregabalin or oxycodone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pain Assessment Training | 1 year
  To assess the ability of Evoked Pain Training (EPT) and Drug/ Placebo Administration (DPA) training to increase subjects' ability to discriminate between active and placebo treatments in a double-blind crossover trial of a known analgesic, measured by standardized effect size, relative to untrained control subjects

SECONDARY OUTCOMES:
Predicted Response to Training | 1 year
  To evaluate whether baseline characteristics of subjects predict response to training, measured by differences in psychophysical profile between baseline and end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wright, MD, Principal Investigator — Analgesic Solutions
Locations (1):
- Analgesic Solutions, Natick, Massachusetts, United States